CLINICAL TRIAL: NCT04218994
Title: The Effect of Instructed Dental Flossing on Interdental Gingival Bleeding: A Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Paul Levi, Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12560
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Gingival Inflammation
Keywords: flossing
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Subjects instructed on flossing technique.
  Interventions: Other: Flossing technique
- Group B (No Intervention): No instructions for flossing provided. Subjects asked to continue their normal oral hygiene care.

INTERVENTIONS:
Other: Flossing technique — Subjects instructed on flossing technique
  Arms: Group A

SUMMARY:
In this study, half of the participants will be asked to floss as normal, while the other half will receive professional instructions on flossing from a dentist. The investigators want to see if the participants who have professional flossing instructions are able to remove plaque in between the teeth more effectively, and have less gum bleeding over time. The investigators also want to see if participants who receive professional flossing instructions get better at the technique over time, and if they can match the dentist's skill by the end of the study.

DETAILED DESCRIPTION:
Primary Aim: To determine whether subjects instructed with a specific flossing technique have less gingival inflammation as evidenced by bleeding on probing (BoP) than subjects without flossing instructions.

Secondary Aim: To compare the effect of flossing by a dental professional with a patient's self-flossing following instruction in removing interdental plaque.

Secondary Aim: To compare the completeness of plaque removal by the subjects instructed during the initial visit (Group A [test]) with their completeness at the final (fourth) visit.

Secondary Aim: To compare the clinician's completeness of plaque removal at the fourth visit with the completeness of plaque removal by the subjects in both groups (Groups A [test] and B [control]). Each group will be analyzed separately. In Group A, a comparison of the plaque removal by the subjects and by the clinician will made with respect to the completeness at the first visit versus the final visit.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Subjects must show > 20% interproximal sites (mesial facial and mesial lingual and distal facial and distal lingual) with BoP. This includes mesial and distal sites next to edentulous areas.
* Subjects must have > 24 natural teeth including teeth with crowns with margins confluent with the natural tooth as long as they do not violate the biologic width.
* Third molars will be excluded from study; unless the third molars are in the anatomical position of second molars. However, subjects with third molars present will be accepted into the study unless there are other factors that exclude them.
* Subjects must report having had a professional dental prophylaxis within four months of beginning the study.
* Subjects must be willing to floss daily and to be taught and use a specific technique of flossing.

Exclusion Criteria:

* Subjects who use tobacco products.
* Subjects with fixed or removable orthodontic appliances
* Subjects with splinted fixed prostheses.
* Subjects who are incapable of flossing their teeth
* Subjects with defective interproximal restorations or interproximal caries that are clinically evident and impacting gingival health.
* Subjects where malposed teeth preclude the use of floss
* Subjects with probing depth greater than or equal to 5mm.
* Subjects who are pregnant (self-reported) due to the greater bleeding tendency due to the hormonal changes.
* Subjects with a systemic disease that affects the gingiva or are taking medications of which affect the gingiva.
* Non-English speaking subjects, as study assessments and instructions will be in English only. There is no direct benefit to subjects for taking part in this study, therefore the exclusion of non-English speaking subjects is not an ethical concern.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Gingival Bleeding Index | Change from Baseline to 8-Week Visit
  The examiner gently swiped the probe at the most apical portion of the gingival crevice from line angle to line angle interproximally and after 10 seconds assessed if there was bleeding or no bleeding on the mesial (facial and lingual) and the distal (facial and lingual).

SECONDARY OUTCOMES:
Modified O'Leary Plaque Score Index | Change from Baseline to 8-Week Visit
  The subjects chewed a Sunstar Butler GUM™ disclosing tablet, and once dissolved in the saliva they swished it in their mouth for 30 seconds. Then they expectorated and rinsed their mouth with water. A plaque index (Modified O'Leary Plaque Score Index Chart) was recorded in which the all teeth surface are stained using a plaque disclosing dye. Plaque was marked as whether present or absent interproximally only for each tooth (buccal and lingual surfaces).
Gingival Bleeding Index | Change from Baseline to 2-Week Visit
  The examiner gently swiped the probe at the most apical portion of the gingival crevice from line angle to line angle interproximally and after 10 seconds assessed if there was bleeding or no bleeding on the mesial (facial and lingual) and the distal (facial and lingual).
Gingival Bleeding Index | Change from Baseline to 4-Week Visit
  The examiner gently swiped the probe at the most apical portion of the gingival crevice from line angle to line angle interproximally and after 10 seconds assessed if there was bleeding or no bleeding on the mesial (facial and lingual) and the distal (facial and lingual).

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States